CLINICAL TRIAL: NCT04615715
Title: Prenatal Behavioral Intervention to Prevent Maternal Cytomegalovirus (CMV) in Pregnancy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Karen Fowler, Primary Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB-300004979; R01HD098352 (NIH)
Record Dates: First submitted 2020-10-21; First posted 2020-11-04 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-10

CONDITIONS: Maternal Cytomegalovirus Infections; Cytomegalovirus Congenital
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Laboratory personnel will not know the participant's intervention status.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CMV Risk-Reduction Intervention (Experimental): One-on-one CMV prevention and education visit followed by 12 weeks of CMV prevention and education text messages
  Interventions: Behavioral: CMV Risk-Reduction Intervention
- Stress Reduction Messaging (Placebo Comparator): One-on-one stress reduction messaging visit followed by 12 weeks of reducing stress text messages
  Interventions: Behavioral: Stress Reduction Messaging

INTERVENTIONS:
Behavioral: CMV Risk-Reduction Intervention — CMV Risk-Reduction Intervention
  Arms: CMV Risk-Reduction Intervention
Behavioral: Stress Reduction Messaging — Stress Reduction Messaging
  Arms: Stress Reduction Messaging

SUMMARY:
This study will evaluate whether a brief prenatal clinic-based cytomegalovirus (CMV) risk-reduction behavioral intervention will prevent maternal CMV infections during pregnancy in women.

DETAILED DESCRIPTION:
Pregnant women will be recruited into the study following their first prenatal visit. After enrollment, they will be randomized to either the CMV risk-reduction intervention or an attention-matched control stress-reduction group stratified by their CMV serostatus.

Women in both groups will attend an individualized behavioral skills session, watch a short video, receive a take-home packet, receive weekly text messages for 12 weeks that reinforce the experimental and control health messages, and attend follow-up visits at 6 and 12 weeks. Saliva, urine, vaginal, and blood specimens will be collected at enrollment and 6 and 12 weeks follow-up visits. Additionally, at-home saliva and vaginal specimen collection will occur at 3 and 9 weeks and once during the third trimester of pregnancy. At delivery, a saliva specimen will be collected from both the mother and infant, along with a remnant cord blood specimen.

ELIGIBILITY:
Inclusion Criteria:

* enrollment in prenatal care before 20 weeks gestation
* absence of CMV IgG on serological testing indicating CMV seronegative status or CMV positive (nonprimary) defined as maternal CMV infection pre-dating pregnancy defined by a high IgG avidity index or a positive CMV IgG in the presence of a negative CMV immunoglobulin M (IgM)

Exclusion Criteria:

* known major fetal anomalies or demise
* planned termination of pregnancy
* planned use of immune globulin, ganciclovir, or valganciclovir
* maternal immune impairment (e.g., HIV infection, organ transplant on anti-rejection medications)
* pre-enrollment ultrasound suggestive of established fetal CMV infection or positive fetal CMV results from culture or PCR
* pre-enrollment CMV seroconversion or primary CMV infection in pregnancy
* unable to determine if CMV infection is a nonprimary infection due to intermediate or undefined CMV serological test results
* pre-enrollment blood, ultrasound, or amniotic fluid testing indicating congenital infection with rubella, syphilis, varicella, parvovirus, toxoplasmosis or other congenital infection
* intention of the patient or of the managing obstetricians for the delivery to be outside of the University of Alabama at Birmingham hospital

Ages: 14 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 840 (Estimated)
Dates: Start 2021-01-11 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
CMV seroconversion rate in CMV seronegative women | Enrollment (baseline) until delivery, up to 32 weeks
  CMV seroconversion is defined as the development of CMV immunoglobulin G (IgG) antibody in the serum of women who did not have antibodies previously. The CMV seroconversion rate will be assessed in participants.
CMV reinfections in women with non-primary infections | Enrollment(baseline) until delivery, up to 32 weeks
  Reinfection will be defined by a combination of strain-specific serologic assays, next-generation sequencing, and virus shedding. The number of CMV reinfections will be assessed in participants.

SECONDARY OUTCOMES:
Change in self-reported CMV risk behaviors and protective behaviors | Enrollment (baseline) to 12 weeks after enrollment (follow-up)
  Change in the CMV risk behaviors and protective behaviors self-reported on the CMV risk behaviors questionnaire at 12 weeks post intervention.
Frequency of CMV shedding | Enrollment(baseline) until delivery, up to 32 weeks
  Number of participants shedding CMV in their specimens collected during pregnancy. CMV shedding is indicated by the presence of CMV DNA by polymerase chain reaction assay (PCR) in saliva, urine, vaginal, or blood specimens.
Proportion of infants with congenital CMV | Delivery
  The proportion of infants with a positive saliva PCR test for CMV in the first 21 days of life.
Frequency of new CMV variants | Enrollment(baseline) until delivery up to 32 weeks
  Number of participants with new CMV variants identified by a combination of serological screening assays and next generation sequencing of viral DNA.

OTHER OUTCOMES:
CMV viral loads | Enrollment(baseline) until delivery, up to 32 weeks
  CMV viral loads indicated by the quantity of CMV DNA by PCR in saliva, urine, vaginal, or blood specimens.
Risk factors for CMV infections | Enrollment(baseline) to 12 weeks after enrollment (follow-up)
  Identification of possible CMV exposures during pregnancy through self-reported exposure questionnaires given at baseline, 6 weeks, and 12 weeks.
Change in anxiety after intervention | Enrollment(baseline) to 12 weeks after enrollment (follow-up)
  Changes in anxiety measured by the Kessler-10 Psychological Distress Scale (K10) administered pre- and post-intervention. K10 scores range from 10 to 50, with 50 indicating highest risk of anxiety.
Change in CMV knowledge | Enrollment(baseline) to 12 weeks after enrollment (follow-up)
  Change in CMV knowledge indicated by self-report on CMV knowledge questionnaire administered pre- and post-intervention to all participants. The questionnaire will be assigned a score of 0 -18 based on the participants' answers, with a higher score indicating desired CMV knowledge.
Acceptability of the educational intervention | Enrollment(baseline) to 12 weeks after enrollment (follow-up)
  Acceptability of prevention messages measured post-intervention by a study assessment questionnaire that provides participant feedback and rating of the intervention at 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Karen B Fowler, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
Requests for data sharing may be considered on a case-by-case basis.